CLINICAL TRIAL: NCT02227303
Title: A Pilot Open Label Clinical Trial to Evaluate the Combined Impact of Two Mobile Health Products on Health Outcomes in Overweight Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medidata Solutions (Industry)
Collaborators: Miami Research Associates (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOVE-2014
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Other)
  Interventions: Behavioral: lifestyle modification instructional and motivational sessions

INTERVENTIONS:
Behavioral: lifestyle modification instructional and motivational sessions

SUMMARY:
The purpose of this study is to explore the effect of 8-weeks use of the Medidata Patient Cloud (a mobile application for capturing data directly from subjects, enabling entry of diary and quality of life data into internet-enabled devices) in combination with an activity tracker (Fitbit Flex) on health outcomes in overweight people with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, aged 18 to 60 years, who are English or Spanish speakers.
2. BMI 25 to 34.9 kg/m2
3. Subject has type 2 diabetes with HgbA1c < 8.0%
4. Subject's glucose is controlled with either diet alone or oral agents that do not cause hypoglycemia (e.g. Metformin, DPP-4 inhibitors, Thiazolidinediones, Alpha-Glucosidase Inhibitors and GLP-1 agonists).
5. Subject is motivated to increase their activity and make other lifestyle changes.
6. Subject has:

   * A compatible Apple mobile device with the iOS 7 operating system installed:

     * iPhone 4 or newer
     * iPad 2 or newer
     * iPad Mini
     * iPod touch 5th gen (2012 model) or newer
   * 500MB of free space on the iPhone, iPad, or iPod touch
   * A valid mobile phone number to receive daily updates via SMS text messaging
   * An active iTunes account/password to install study-related software ("apps")
   * Access to Wi-Fi or a mobile data plan to send study data
7. Female subject is surgically sterile, post-menopausal or agrees to use an acceptable method of birth control as defined in section 2.7.
8. Subject agrees to not use any new vitamin and/or mineral supplement until after study completion.
9. Subject agrees to not take any dietary or herbal supplements or products until after study completion. Seven-day washout period prior to study inclusion allowed.
10. Subject is willing and able to comply with the protocol including:

    1. Attending 3 visits, approximately 2 hours each
    2. Wearing and inputting required information into the Fitbit Flex activity tracker
    3. Receiving alerts from the Medidata Patient Cloud
    4. Working on making nutrition and exercise changes over the 8-week study period
    5. Using and updating his/her iPhone, iPad, iPad Mini or iTouch as per study requirements (e.g. downloading the iOS7 operating system, downloading the Medidata Patient Cloud and Fitbit Flex apps, and receiving daily text messages).
11. Subject is able to understand and sign the informed consent to participate in the study.

Exclusion Criteria:

1. Subject has any of the following medical conditions:

   1. active heart disease
   2. uncontrolled high blood pressure (≥ 140/90 mmHg)
   3. renal or hepatic impairment/disease
   4. Type I diabetes
   5. bipolar disorder
   6. active psychiatric disease
   7. Parkinson's disease
   8. unstable thyroid disease
   9. immune disorder (such as HIV/AIDS)
   10. any medical condition deemed exclusionary by the Principal Investigator (PI)
2. Subject has a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within five years prior to screening.
3. Subject is taking oral agents that can cause hypoglycemia (e.g. sulfonylureas, meglitinides and insulin).
4. Subject is taking or has taken in the past 28 days any supplement or medication (prescription or over the counter) for weight loss (see section 2.6.2); 28-day washout required for study inclusion.
5. Subject is on an unstable dose of medication (defined as fewer than 90 days at the same dose).
6. Subject is currently taking any medication deemed exclusionary by PI.
7. Subject exhibits evidence of hepatic or renal dysfunction as evidenced by ALT, AST, AP being ≥ 2 times the upper limit of normal or serum creatinine value ≥ 2.0 mg/dl or other clinically significant abnormal clinical laboratory value per PI discretion.
8. Subject has a clinically relevant abnormality as defined by the PI or interpreting physician with respect to the electrocardiogram (ECG).
9. Subject has a QTc interval > 450 msec for males and > 470 msec for females.
10. Subject has a history of drug or alcohol abuse in the past 12 months.
11. Subject has begun/stopped smoking ≤ 6 months ago OR has plans to begin/quit smoking.
12. Subject has experienced a weight loss or gain greater than 4.5 kg (approximately 10 lbs) in the past 3 months.
13. Subject is pregnant, lactating, or planning to become pregnant during the study period.
14. Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
15. Subject has taken an investigational product within 30 days of study enrollment (visit 2).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to 8 weeks in glucose, insulin, fructosamine and HgbA1c | 8 weeks
Changes from baseline to 4 and 8 weeks in body weight. | 4 to 8 weeks
Changes from baseline to 4 and 8 weeks in compliance with nutrition goals as measured via dichotomous questionnaire. | 4 to 8 weeks
Changes from baseline to 4 and 8 weeks in compliance with exercise goals as measured by steps per day (provided by the Fitbit Flex). | 4 to 8 weeks
Weekly changes over 8 weeks as compared to baseline in quality of life as measured by the PROMIS® Global Health questionnaire (global physical health and global mental health subscale scores and social and overall health scores). | 8 weeks

OTHER OUTCOMES:
Changes from baseline to 4 and 8 weeks on quality of sleep as measured via the sleep efficiency score (provided by the Fitbit Flex). | 4 to 8 weeks
Changes from baseline to 4 and 8 weeks in compliance with exercise goals as measured by active minutes (provided by the Fitbit Flex; requires subject input of data). | 4 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane R. Krieger, MD, Principal Investigator — Miami Research Associates. Miami, FL.
Locations (1):
- Miami Research Associates (MRA), Miami, Florida, United States

REFERENCES:
- [Background] Evert AB, Boucher JL, Cypress M, Dunbar SA, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Nwankwo R, Verdi CL, Urbanski P, Yancy WS Jr. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes Care. 2014 Jan;37 Suppl 1:S120-43. doi: 10.2337/dc14-S120. No abstract available. PMID 24357208
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343